CLINICAL TRIAL: NCT05414318
Title: Post Marketing Surveillance of the Conformable GORE® TAG® Thoracic Endoprosthesis (CTAG)
Brief Title: CTAG Dissection/Trauma Post Marketing Surveillance Japan
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 16-01
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Aortic Aneurysm; Thoracic Aorta Injury; Thoracic Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Conformable GORE® TAG® Thoracic Endoprosthesis — Thoracic Endoprosthesis

SUMMARY:
Post Marketing Surveillance of the Conformable GORE® TAG® Thoracic Endoprosthesis

ELIGIBILITY:
Inclusion Criteria for Acute, Complicated Stanford Type B Aortic Dissection:

* Patient present with acute complicated type B aortic dissection
* Patient who do not respond to medical therapy
* Time from symptom onset to dissection diagnosis ≤ 14 days
* Adequate iliac / femoral access or conduit
* Aortic inner diameter at proximal extent of proximal landing zone in the range of 16-42 mm
* ≥ 20 mm landing zone proximal to the primary entry tear; proximal extent of the landing zone must not be dissected

Inclusion Criteria for Traumatic Aortic Transection:

* Patient has traumatic aortic transection that requires repair as determined by treating physician
* Adequate iliac / femoral access
* Aortic inner diameter in the range of 16-42 mm on the proximal and distal sides
* ≥ 20 mm non-aneurysmal aorta neck proximal and distal to the lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute, complicated Stanford Type B aortic dissection and patients with traumatic aortic transection treated using Gore CTAG.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Dissection: Acute complicated Stanford type B dissection: Patients are enrolled and surveyed if the device is used in patients with complicated acute Stanford Type B aortic dissection at sites that contracted for this survey
- Trauma: Traumatic thoracic aortic injury: Patients are enrolled and surveyed if the device is used in patients with Traumatic thoracic aortic injury at sites that contracted for this survey
Period: Overall Study
Arm/Group | Dissection | Trauma
Started | 43 | 12
Completed | 21 | 5
Not Completed | 22 | 7

BASELINE CHARACTERISTICS:
Groups:
- Dissection: Acute complicated Stanford type B dissection
- Trauma: Traumatic thoracic aortic injury
- Total: Total of all reporting groups
Arm/Group | Dissection | Trauma | Total
Number analyzed (Participants) | 43 | 12 | 55
Age, Continuous [Median (Full Range); unit: years] — Population: Missing Data for Some Participants
  years
    number analyzed (Participants) | 38 | 12 | 50
    (all) | 65 [40 to 89] | 58.5 [20 to 79] | 65 [20 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 33 | 10 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 43 | 12 | 55
Height [Median (Full Range); unit: cm] — Population: Missing Data for Some Participants
  cm
    number analyzed (Participants) | 38 | 10 | 48
    (all) | 165 [145 to 180] | 166.5 [155 to 182] | 165 [145 to 182]
Weight [Median (Full Range); unit: kg] — Population: Missing Data for Some Participants
  kg
    number analyzed (Participants) | 41 | 12 | 53
    (all) | 63.9 [30.3 to 94.8] | 67.3 [47.3 to 98.0] | 66.0 [30.3 to 98.0]
American Society of Anesthesiologists (ASA) Classification [Count of Participants; unit: Participants] — ASA I - Healthy patient for elective operation ASA II - Patient with mild systemic disease limits activity but is not incapacitating ASA III - Patient with severe systemic disease that is constant threat of life, limits activity but is not incapacitating ASA IV - Patient with incapacitating disease that is a constant threat of life ASA V - Moribund patient not expected to live 24 hours with or without operation
  Participants
    ASA 1 | 13 | 3 | 16
    ASA II | 10 | 0 | 10
    ASA III | 11 | 5 | 16
    ASA IV | 9 | 4 | 13
    ASA V | 0 | 0 | 0
Pulmonary Disease [Count of Participants; unit: Participants] | 4 | 0 | 4
Renal Disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Cerebrovascular Disease [Count of Participants; unit: Participants] | 6 | 0 | 6
Hypertension [Count of Participants; unit: Participants] | 29 | 2 | 31
Diabetes Mellitus [Count of Participants; unit: Participants] | 5 | 1 | 6
Prior Descending Thoracic Aorta Repair [Count of Participants; unit: Participants] | 0 | 0 | 0
At Risk for Graft Infection [Count of Participants; unit: Participants] | 0 | 1 | 1
Persistent Refractory Shock [Count of Participants; unit: Participants] | 3 | 2 | 5
Bowel Necrosis [Count of Participants; unit: Participants] | 1 | 0 | 1
Degenerative Connective Tissue Disease [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Entry Tear Exclusion
Description: Number of subjects who achieved the primary entry tear exclusion
Time Frame: At each follow-up visit through 5 years: 1 Month (15-59 days), 6 Months (60-242 days), 12 Months (243-546 days), 24 Months (547-911 days), 36 Months (912-1275 days), 48 Months (1276-1640 days), 60 Months (1641-2006 days)
Population: Patients with acute complicated Stanford type B dissection with evaluable result. (Not a protocol-defined endpoint for trauma arm and therefore not evaluated)
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection
Number analyzed (Participants) | 38
Participants
  1 Month: number analyzed (Participants) | 23
  1 Month | 21
  6 Months: number analyzed (Participants) | 26
  6 Months | 26
  12 Months: number analyzed (Participants) | 27
  12 Months | 27
  24 Months: number analyzed (Participants) | 23
  24 Months | 22
  36 Months: number analyzed (Participants) | 19
  36 Months | 19
  48 Months: number analyzed (Participants) | 17
  48 Months | 17
  60 Months: number analyzed (Participants) | 20
  60 Months | 20

2. Primary Outcome: Aortic Rupture
Description: Number of subjects with Aortic Rupture
Time Frame: Procedure through 5 years (Day 0-2006)
Population: Subjects with acute complicated Stanford type B dissection. (Not a protocol-defined endpoint for trauma arm and therefore not evaluated)
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection
Number analyzed (Participants) | 43
Participants | 2

3. Primary Outcome: Major Device-related Adverse Events
Description: Number of subjects with major device-related adverse events
Time Frame: Procedure through 5 years (Day 0-2006)
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection | Trauma
Number analyzed (Participants) | 43 | 12
Participants | 3 | 0

4. Primary Outcome: Secondary Intervention Treatment
Description: Incidence rate of secondary intervention treatment
Time Frame: Post-procedure through 5 years (Day 1-2006)
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection | Trauma
Number analyzed (Participants) | 42 | 12
Participants | 5 | 0

5. Primary Outcome: Change in Minimum True Lumen Diameter Adjacent to Treated Segment
Description: Change in minimum true lumen diameter adjacent to treated segment at each follow-up visit:
  Decrease (>=5mm) vs No change vs Increase (>=5mm)
Time Frame: as for outcome 1
Population: Patients with acute complicated Stanford type B dissection with evaluable result. (Outcome not applicable for trauma arm - see Outcome Measure #9 for change in maximum lesion diameter for the trauma arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection
Number analyzed (Participants) | 38
Participants
  1 Month: number analyzed (Participants) | 25
  1 Month: Decrease | 1
  1 Month: No Change | 6
  1 Month: Increase | 18
  6 Months: number analyzed (Participants) | 30
  6 Months: Decrease | 1
  6 Months: No Change | 3
  6 Months: Increase | 26
  12 Months: number analyzed (Participants) | 31
  12 Months: Decrease | 0
  12 Months: No Change | 7
  12 Months: Increase | 24
  24 Months: number analyzed (Participants) | 29
  24 Months: Decrease | 0
  24 Months: No Change | 6
  24 Months: Increase | 23
  36 Months: number analyzed (Participants) | 22
  36 Months: Decrease | 0
  36 Months: No Change | 4
  36 Months: Increase | 18
  48 Months: number analyzed (Participants) | 19
  48 Months: Decrease | 0
  48 Months: No Change | 3
  48 Months: Increase | 16
  60 Months: number analyzed (Participants) | 21
  60 Months: Decrease | 0
  60 Months: No Change | 3
  60 Months: Increase | 18

6. Primary Outcome: Change in Minimum True Lumen Diameter Distal to Treated Segment
Description: Change in minimum true lumen diameter distal to treated segment at each follow-up visit:
  Decrease (>=5mm) vs No change vs Increase (>=5mm)
Time Frame: as for outcome 1
Population: Patients with acute complicated Stanford type B dissection with evaluable result (Outcome not applicable for trauma arm - see Outcome Measure #9 for change in maximum lesion diameter for the trauma arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection
Number analyzed (Participants) | 37
Participants
  1 Month: number analyzed (Participants) | 24
  1 Month: Decrease | 0
  1 Month: No Change | 13
  1 Month: Increase | 11
  6 Months: number analyzed (Participants) | 26
  6 Months: Decrease | 1
  6 Months: No Change | 11
  6 Months: Increase | 14
  12 Months: number analyzed (Participants) | 26
  12 Months: Decrease | 0
  12 Months: No Change | 10
  12 Months: Increase | 16
  24 Months: number analyzed (Participants) | 26
  24 Months: Decrease | 0
  24 Months: No Change | 7
  24 Months: Increase | 19
  36 Months: number analyzed (Participants) | 20
  36 Months: Decrease | 0
  36 Months: No Change | 5
  36 Months: Increase | 15
  48 Months: number analyzed (Participants) | 18
  48 Months: Decrease | 0
  48 Months: No Change | 6
  48 Months: Increase | 12
  60 Months: number analyzed (Participants) | 20
  60 Months: Decrease | 0
  60 Months: No Change | 7
  60 Months: Increase | 13

7. Primary Outcome: Change in Maximum False Lumen Diameter Adjacent to Treated Segment
Description: Change in maximum false lumen diameter adjacent to treated segment at each follow-up visit:
  Decrease (>=5mm) vs No change vs Increase (>=5mm)
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection
Number analyzed (Participants) | 38
Participants
  1 Month: number analyzed (Participants) | 24
  1 Month: Decrease | 18
  1 Month: No Change | 5
  1 Month: Increase | 1
  6 Months: number analyzed (Participants) | 27
  6 Months: Decrease | 23
  6 Months: No Change | 4
  6 Months: Increase | 0
  12 Months: number analyzed (Participants) | 29
  12 Months: Decrease | 24
  12 Months: No Change | 4
  12 Months: Increase | 1
  24 Months: number analyzed (Participants) | 25
  24 Months: Decrease | 21
  24 Months: No Change | 2
  24 Months: Increase | 2
  36 Months: number analyzed (Participants) | 20
  36 Months: Decrease | 17
  36 Months: No Change | 2
  36 Months: Increase | 1
  48 Months: number analyzed (Participants) | 18
  48 Months: Decrease | 15
  48 Months: No Change | 2
  48 Months: Increase | 1
  60 Months: number analyzed (Participants) | 19
  60 Months: Decrease | 18
  60 Months: No Change | 0
  60 Months: Increase | 1

8. Primary Outcome: Change in Maximum False Lumen Diameter Distal to Treated Segment
Description: Change in maximum false lumen diameter distal to treated segment at each follow-up visit:
  Decrease (>=5mm) vs No change vs Increase (>=5mm)
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Dissection
Number analyzed (Participants) | 37
Participants
  1 Month: number analyzed (Participants) | 24
  1 Month: Decrease | 14
  1 Month: No Change | 10
  1 Month: Increase | 0
  6 Months: number analyzed (Participants) | 25
  6 Months: Decrease | 19
  6 Months: No Change | 5
  6 Months: Increase | 1
  12 Months: number analyzed (Participants) | 26
  12 Months: Decrease | 20
  12 Months: No Change | 4
  12 Months: Increase | 2
  24 Months: number analyzed (Participants) | 23
  24 Months: Decrease | 15
  24 Months: No Change | 6
  24 Months: Increase | 2
  36 Months: number analyzed (Participants) | 19
  36 Months: Decrease | 12
  36 Months: No Change | 3
  36 Months: Increase | 4
  48 Months: number analyzed (Participants) | 17
  48 Months: Decrease | 14
  48 Months: No Change | 1
  48 Months: Increase | 2
  60 Months: number analyzed (Participants) | 19
  60 Months: Decrease | 15
  60 Months: No Change | 3
  60 Months: Increase | 1

9. Primary Outcome: Change in Maximum Lesion Diameter
Description: Change in maximum lesion diameter at each follow-up visit:
  Decrease (>=5mm) vs No change vs Increase (>=5mm)
Time Frame: At each follow-up visit from 6 months through 5 years: 6 Months (60-242 days), 12 Months (243-546 days), 24 Months (547-911 days), 36 Months (912-1275 days), 48 Months (1276-1640 days), 60 Months (1641-2006 days)
Population: Subjects with Traumatic thoracic aortic injury. (Outcome not applicable for dissection arm - see Outcome Measures #5-8 for change in true/false lumen diameter for the dissection arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Trauma
Number analyzed (Participants) | 3
Participants
  6 Months: Decrease | 1
  6 Months: No Change | 2
  6 Months: Increase | 0
  12 Months: Decrease | 1
  12 Months: No Change | 2
  12 Months: Increase | 0
  24 Months: Decrease | 1
  24 Months: No Change | 2
  24 Months: Increase | 0
  36 Months: number analyzed (Participants) | 1
  36 Months: Decrease | 1
  36 Months: No Change | 0
  36 Months: Increase | 0
  48 Months: number analyzed (Participants) | 2
  48 Months: Decrease | 1
  48 Months: No Change | 1
  48 Months: Increase | 0
  60 Months: number analyzed (Participants) | 1
  60 Months: Decrease | 1
  60 Months: No Change | 0
  60 Months: Increase | 0

ADVERSE EVENTS:
Time Frame: 5 years (Post-operative day 0-2006)
Arm/Group | Dissection | Trauma
All-Cause Mortality (participants affected / at risk) | 10/43 | 1/12
Serious Adverse Events (participants affected / at risk) | 17/43 | 1/12
Other Adverse Events (participants affected / at risk) | 0/43 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dissection (N=43) | Trauma (N=12)
Aortic Rupture (Vascular disorders) | 2 | 0
New Aortic Dissection (Vascular disorders) | 2 | 0
False Lumen Enlargement (>=5mm) (Vascular disorders) | 1 | 0
Atelactasis/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Congestive Heart Failure (Cardiac disorders) | 3 | 0
Bowel Ischemia (Gastrointestinal disorders) | 3 | 0
Other Bowel Complication (Gastrointestinal disorders) | 1 | 0
Other Vascular Complication (Vascular disorders) | 1 | 0
Paraplegia/Paraparesis (Nervous system disorders) | 1 | 0
Prosthesis Infection (Infections and infestations) | 2 | 0
Other Infection (Infections and infestations) | 1 | 0
Other Complications (not device complication) (General disorders) | 3 | 1
Endoleak Type Ia (Vascular disorders) | 1 | 0
Endoleak Type III (Vascular disorders) | 1 | 0
Endoleak, Other (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is required to obtain written permission from the Sponsor prior to publishing trial results.

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT05414318/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT05414318/SAP_001.pdf